CLINICAL TRIAL: NCT02814903
Title: ALDOsterone for Prediction of Post-Operative Atrial Fibrillation
Acronym: ALDO-POAF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: A14-D05-VOL.20
Record Dates: First submitted 2016-06-14; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Atrial Fibrillation
Keywords: aldosterone; cardiac surgery; atrial fibrillation; galectin-3; mitochondria; ngal; acute kidney failure; epicardial fat; right atrial sample
MeSH Terms: conditions — Atrial Fibrillation; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — * aldosterone
  * galectin 3
  * ngal
  * mitochondria
  * right atrial sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Planned cardiac surgery. POAF occurence or not: The ALDO-POAF study is an observational, 1-center and prospective pilot study that will enroll patients undergoing CABG ± aortic valve replacement. Patients who had emergency CABG, need for concomitant mitral surgery, left ventricular ejection fraction (LVEF) < 50%, a history of AF or other atrial arrhythmia, unstable angina or heart failure, cardiogenic shock, atrioventricular block, hypothyroidism/hyperthyroidism, previous heart surgery, and off-pump or on-pump beating CABG will be excluded.

SUMMARY:
Post-operative atrial fibrillation (POAF) is a major and frequent complication occurring after cardiac surgery, contributing to prolonged intensive care and hospital stays and is associated with several cardiovascular complications. The exact mechanisms and signaling pathways involved in the development of POAF seem to be multifactorial and remain to date incompletely understood. β-blockers and amiodarone are the first line preventive drugs but are partially effective and near 30% of POAF resist to these strategies. In this context, there is some evidence indicating that renin-angiotensin-aldosterone system and Galectin-3 (Gal-3) share signaling pathways in the development of cardiac fibrosis and therefore could be very useful predictive biomarkers of POAF and potentially interesting therapeutic target to prevent POAF occurrence.

The investigators hypothesis is that preoperative plasma aldosterone levels and galectin-3 (Gal-3) expression (in plasma, right atrial appendage or epicardial fat) could be predictive of POAF in patients undergoing elective CABG surgery with preserved LVEF.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for planned surgical coronary revascularization +/- aortic replacement valve
* Aged 18 years at least
* Clinically Stable (see criteria for non-inclusion)
* With left ventricular ejection fraction preserved (>50%)

Exclusion Criteria:

* Patient having already AF history
* Patient with primary hyperaldosteronism
* Unstable Patient defined as any cardiovascular event occurred in the previous 30 days

These events are:

* hospitalisation for cardiovascular causes
* appearance or worsening of symptoms consistent with cardiac failure
* appearance or worsening symptoms of coronary
* Patient refusing participation in the study
* Patient unable to provide follow-up visits
* need for concomitant mitral surgery
* Emergency CABG
* Left ventricular ejection fraction (LVEF) < 50%
* Previous heart surgery
* Off pump CABG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The ALDO-POAF study is an observational, 1-center and prospective pilot study that will enroll patients undergoing CABG ± aortic valve replacement. Patients who had emergency CABG, need for concomitant mitral surgery, left ventricular ejection fraction (LVEF) < 50%, a history of AF or other atrial arrhythmia, unstable angina or heart failure, cardiogenic shock, atrioventricular block, hypothyroidism/hyperthyroidism, previous heart surgery, and off-pump or on-pump beating CABG will be excluded. Approval for this study, including collection of human tissues (right atrial appendage, subcutaneous and epicardial fat) and blood collection, was obtained from the Ethics Committee of Caen University Hospital (Comité de Protection des Personnes Nord-Ouest III, Caen, France) and will be in accordance to the declaration of Helsinki; the details of the study will be explained to the subjects, and written informed consent will be obtained from each patient.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Occurrence of atrial fibrillation in post-operative period of cardiac surgery (CABG +/- aortic valve replacement) | 1 month

SECONDARY OUTCOMES:
Find a correlation between the local secretion of aldosterone by adipocytes epicardial and the occurrence of AF during the 6 months after surgery in patients undergoing cold bypass coronary artery. | 6 months
Find a correlation between aldosterone levels secreted in epicardial adipocytes and plasma aldosterone levels. | 1 month
Find a correlation between preoperative plamastic aldosterone levels and occurence of postoperative atrial fibrillation | 1 month
Detect aldosterone synthase aldosterone or angiotensin II (measured by quantitative and qualitative assays Western Blot, mRNA or RT-PCR) in the epicardial fat removed during surgery in patients undergoing a CABG. | 1 month
Find a correlation between preoperative plamastic galectin-3 levels and occurrence of postoperative atrial fibrillation | 1 month
Find a correlation between preoperative plamastic ngal levels and occurrence of postoperative atrial fibrillation | 1 month
Find a correlation between preoperative mitochondrial function and occurrence of postoperative atrial fibrillation | 1 month
Find a correlation between preoperative left atrial strain and occurrence of postoperative atrial fibrillation | 1 month
Find a correlation between acute renal failure and occurrence of postoperative atrial fibrillation | 1 month
Find a correlation between occurrence of postoperative atrial fibrillation and all cause cardiovascular morbimortality | 2 years
Find a correlation between occurrence of postoperative atrial fibrillation and length of hospitalisation | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Joachim ALEXANDRE, Caen, Basse Normandie, France

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ollitrault P, Allouche S, Chequel M, Milliez P, Alexandre J. Plasma aldosterone and atrial mitochondrial functions of patients undergoing cardiac surgery. Future Cardiol. 2020 Jul;16(4):275-280. doi: 10.2217/fca-2019-0028. Epub 2020 Apr 14. PMID 32286862